CLINICAL TRIAL: NCT03462381
Title: The Impact of Protein Supplementation to Maximize Skeletal Muscle Endurance Training Adaptations in Healthy Young Men
Brief Title: Protein Supplementation and Endurance Exercise Adaptations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NL5988508116
Record Dates: First submitted 2017-09-26; First posted 2018-03-12 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity | interventions — Proteins

STUDY DESIGN:
Intervention Model Description: Participants will perform three endurance training sessions weekly for 12 weeks. All participants will be randomly assigned to the protein supplementation group or the placebo (iso-caloric carbohydrate) group. During the 12 weeks endurance training program participants allocated to the protein group (30 g protein per beverage) will receive a protein drink after exercise and prior to sleep at night on training days. On non-training days participants will only receive a protein drink before sleep. Participants allocated to the carbohydrate group (30 g carbohydrates) will receive a carbohydrate drink instead of a protein drink.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein (Experimental): Three endurance training sessions weekly with protein supplementation post-exercise and before sleep.
  Interventions: Dietary Supplement: Protein
- Carbohydrate (Placebo Comparator): Three endurance training sessions weekly with carbohydrate supplementation post-exercise and before sleep.
  Interventions: Dietary Supplement: Protein

INTERVENTIONS:
Dietary Supplement: Protein — Three endurance training sessions weekly with protein supplementation post-exercise and before sleep.

SUMMARY:
Participants will perform three endurance training sessions weekly for 12 weeks. All participants will be randomly assigned to the protein supplementation group or the placebo (iso-caloric carbohydrate) group. During the 12 weeks endurance training program participants allocated to the protein group (30 g protein per beverage) will receive a protein drink after exercise and prior to sleep at night on training days. On non-training days participants will only receive a protein drink before sleep. Participants allocated to the carbohydrate group (30 g carbohydrates) will receive a carbohydrate drink instead of a protein drink.

DETAILED DESCRIPTION:
In the proposed study, the effects of protein supplementation after training and before sleep on VO2max and performance will be assessed during 12 weeks endurance exercise training in untrained healthy young men. The ready to drink carbohydrate beverage consists of 30g carbohydrate or 30g protein. Previous studies show that the supplementation of 30g protein is in the optimal range to stimulate the muscle protein synthetic response following resistance type exercise. The protein supplementation group in the present study will be compared with an iso-caloric carbohydrate group. In addition, to the pre- and post-intervention biopsies 1 additional muscle biopsies will be taken (in week 6) during the 12 week intervention period. This will create a unique opportunity to establish the timeline of the skeletal muscle adaptive response at functional and mechanistic level following prolonged endurance exercise training, including potential differences between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 18 and 30 years of age
* BMI between 18.5 - 25 kg/m2
* Recreationally active, performing sports on a non-competitive basis
* Maximal wattage of > 5 watt per kg bodyweight (screening measurement)
* Willing to give muscle biopsies
* Willing to give blood samples
* Having a general-practitioner
* Consumption of alcohol beverages is less than 21 per week
* Able to perform three exercise sessions weekly for 10 weeks

Exclusion Criteria:

* Medical condition that can interfere with the study outcome (i.e. cardiovascular disease, pulmonary disease, liver or renal disease, diabetes mellitus type 1 or 2)
* Having a lactose and/or gluten intolerance
* Use of systemic medication (with the exception of antihistaminic medication and the use of occasional painkillers)
* (Chronic) injuries of the locomotor system (e.g. musculoskeletal/orthopedic disorders) that can interfere with the intervention
* Participants who are enrolled in an interventional biomedical research project or have received an investigational new drug or product with the last 30 days prior to screening.
* Smokers and use of illicit drugs
* Blood donor during the study and in the three months before start of the study
* Employed, or intern, or working on a thesis at the department of Human Nutrition at Wageningen University & Research
* Participating in another scientific study (except EetMeetWeet)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Young healthy men
Enrollment: 44 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Maximal whole-body oxidative capacity | Baseline
  Maximal oxygen consumption in ml per kg of bodyweight
Maximal whole-body oxidative capacity | 6 weeks
  Maximal oxygen consumption in ml per kg of bodyweight
Maximal whole-body oxidative capacity | 12 weeks
  Maximal oxygen consumption in ml per kg of bodyweight

SECONDARY OUTCOMES:
Endurance Performance | Baseline
  10-km simulated time trial performance in seconds
Endurance Performance | 6 weeks
  10-km simulated time trial performance in seconds
Endurance Performance | 12 weeks
  10-km simulated time trial performance in seconds
Maximal activity of citrate synthase | Baseline
  Maximal activity of citrate synthase in micromol per gram per minute
Maximal activity of citrate synthase | 6 weeks
  Maximal activity of citrate synthase in micromol per gram per minute
Maximal activity of citrate synthase | 12 weeks
  Maximal activity of citrate synthase in micromol per gram per minute
Maximal activity of Cytochrome c oxidase | Baseline
  Maximal activity of Cytochrome c oxidase in micromol per gram per minute
Maximal activity of Cytochrome c oxidase | 6 weeks
  Maximal activity of Cytochrome c oxidase in micromol per gram per minute
Maximal activity of Cytochrome c oxidase | 12 weeks
  Maximal activity of Cytochrome c oxidase in micromol per gram per minute
Erythrocytes | Baseline
  Erythrocytes count/pL
Erythrocytes | 2 weeks
  Erythrocytes count/pL
Erythrocytes | 4 weeks
  Erythrocytes count/pL
Erythrocytes | 6 weeks
  Erythrocytes count/pL
Erythrocytes | 8 weeks
  Erythrocytes count/pL
Erythrocytes | 10 weeks
  Erythrocytes count/pL
Erythrocytes | 12 weeks
  Erythrocytes count/pL
Hemoglobin | Baseline
  Hemoglobin mmol/L
Hemoglobin | 2 weeks
  Hemoglobin mmol/L
Hemoglobin | 4 weeks
  Hemoglobin mmol/L
Hemoglobin | 6 weeks
  Hemoglobin mmol/L
Hemoglobin | 8 weeks
  Hemoglobin mmol/L
Hemoglobin | 10 weeks
  Hemoglobin mmol/L
Hemoglobin | 12 weeks
  Hemoglobin mmol/L
Hematocrit | Baseline
  Hematocrit L/L
Hematocrit | 2 weeks
  Hematocrit L/L
Hematocrit | 4 weeks
  Hematocrit L/L
Hematocrit | 6 weeks
  Hematocrit L/L
Hematocrit | 8 weeks
  Hematocrit L/L
Hematocrit | 10 weeks
  Hematocrit L/L
Hematocrit | 12 weeks
  Hematocrit L/L
Lean mass | Baseline
  Lean mass kg
Lean mass | 6 weeks
  Lean mass kg
Lean mass | 12 weeks
  Lean mass kg
Fat mass | Baseline
  Fat mass kg
Fat mass | 6 weeks
  Fat mass kg
Fat mass | 12 weeks
  Fat mass kg

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University & Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knuiman P, Hangelbroek R, Boekschoten M, Hopman M, Mensink M. Impact of protein supplementation during endurance training on changes in skeletal muscle transcriptome. BMC Genomics. 2020 Jun 9;21(1):397. doi: 10.1186/s12864-020-6686-x. PMID 32517654
- [Derived] Knuiman P, van Loon LJC, Wouters J, Hopman M, Mensink M. Protein supplementation elicits greater gains in maximal oxygen uptake capacity and stimulates lean mass accretion during prolonged endurance training: a double-blind randomized controlled trial. Am J Clin Nutr. 2019 Aug 1;110(2):508-518. doi: 10.1093/ajcn/nqz093. PMID 31240303